CLINICAL TRIAL: NCT01127776
Title: APOS System Effects in Post-operation Bi-trimalleolar Fracture of Ankle Prospective, Comparative Randomize Trial Study
Brief Title: Bi-trimalleolar Fracture and APOS System Treatment
Acronym: APOS-IL 001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC9181-09CTIL
Record Dates: First submitted 2010-04-27; First posted 2010-05-21 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Bi-trimalleolar Fracture of Ankle
Keywords: patient after bi-trimalleolar fracture of ankle

ARMS (2):
- Apos System (Experimental)
  Interventions: Device: APOS SYSTEM
- CONTROL (Placebo Comparator)
  Interventions: Other: APOS SYSTEM without biomechanics units.

INTERVENTIONS:
Device: APOS SYSTEM — The trial group will receive APOS walking system The control group will receive the same walking protocol as the trial group without biomechanics units
  Arms: Apos System
Other: APOS SYSTEM without biomechanics units. — The control group will receive the same walking protocol as the trial group without biomechanics units
  Arms: CONTROL

SUMMARY:
The purpose of this study is to evaluate of functional tests and clinical findings with APOS System treatment in patient after bi-trimalleolar fracture of ankle. These functional changes will be evaluated AOFS, FAOS, SF36 and WOMAC scores, walking laboratory GAITRite and clinical examination.

DETAILED DESCRIPTION:
Trial design Prospective, comparative, randomize trial. The patients after surgery due to bi or trimalleolar fracture of ankle, that were referred to the physiotherapy treatment, 3 weeks cast and 6 weeks from surgery with full weight bearing indicated by orthopedic

* The population will randomized separated in trail and control group/ Both receive APOS shoes The trial group will receive APOS walking system
* The control group will receive the same walking protocol as the trial group without biomechanics units.

  1. st visit: enrollment of patient - 6 weeks post op 1. The patient will be given a full verbal and written explanation regarding the trial and treatment. The patient will sign the informed consent form and will be given a serial number.

  2. The screening forms will be completed. 3. Demographic data: date of birth, sex, age and complete medical history, height and previous treatments will be recorded.

  4. Physical examination: range of motion, Achilles tendon thickness. The results will be recorded in the CRF 5. Walking test using a laboratory walking GAITRite + 6 minute walk test 6. Fill out questionnaire: FAOS - AOSF - SF36 - WOMAC 7. Adjustment of Apos walking System

  2nd visit: 12 weeks post op
  1. Physical examination: range of motion, Achilles tendon thickness. The results will be recorded in the CRF
  2. Walking test using a laboratory walking GAITRite + 6 minute walk test
  3. Fill out questionnaire: FAOS - AOSF - SF36 - WOMAC

  3rd visit: 3 month post op
  1. Physical examination: range of motion, Achilles tendon thickness. The results will be recorded in the CRF
  2. Walking test using a laboratory walking GAITRite + 6 minute walk test
  3. Fill out questionnaire: FAOS - AOSF - SF36 - WOMAC

  4th visit: 6 month post op
  1. Physical examination: range of motion, Achilles tendon thickness. The results will be recorded in the CRF
  2. Walking test using a laboratory walking GAITRite + 6 minute walk test
  3. Fill out questionnaire: FAOS - AOSF - SF36 - WOMAC

  5th visit: 12 month post op

  1. Physical examination: range of motion, Achilles tendon thickness. The results will be recorded in the CRF 2. Walking test using a laboratory walking GAITRite + 6 minute walk test 3. Fill out questionnaire: FAOS - AOSF - SF36 - WOMAC

  6th visit: 18 month post op
  1. Physical examination: range of motion, Achilles tendon thickness. The results will be recorded in the CRF
  2. Walking test using a laboratory walking GAITRite + 6 minute walk test
  3. Fill out questionnaire: FAOS - AOSF - SF36 - WOMAC

  7th visit: 24 month post op
  1. Physical examination: range of motion, Achilles tendon thickness. The results will be recorded in the CRF
  2. Walking test using a laboratory walking GAITRite + 6 minute walk test
  3. Fill out questionnaire: FAOS - AOSF - SF36 - WOMAC

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18-65 year old
* Post operation bi- trimalleolar fracture of ankle
* Download cast after 3 weeks
* Full Weight bearing after 6 weeks
* Patients in medical condition to receive physiotherapy treatment
* Patients who are willing to participate in the trial, to come to all scheduled visits and to sign the informed consent forms.

Exclusion Criteria:

* Patients suffering muscular or nerve disorders
* Patients who are unable to use the APOS SYSTEM and can not complete the experimental protocol due to physical or mental handicap
* Non cooperative patient with the basic rehab program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
APOS System effects | one year
  Evaluate with functional tests and clinical findings patient after bi-trimalleolar fracture of ankle with who recive APOS System treatment.
  Functional changes will be evaluated using FAOS, SF36 and WOMAC scores, walking laboratory GAITRite and clinical examination.

SECONDARY OUTCOMES:
Ankle fracture | one year
  bi-trimalleolar ankle fracture - crif

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Department - Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Derived] Lewis SR, Pritchard MW, Parker R, Searle HKC, Beckenkamp PR, Keene DJ, Bretherton C, Lin CC. Rehabilitation for ankle fractures in adults. Cochrane Database Syst Rev. 2024 Sep 23;9(9):CD005595. doi: 10.1002/14651858.CD005595.pub4. PMID 39312389
- [Derived] Segal G, Elbaz A, Parsi A, Heller Z, Palmanovich E, Nyska M, Feldbrin Z, Kish B. Clinical outcomes following ankle fracture: a cross-sectional observational study. J Foot Ankle Res. 2014 Nov 28;7(1):50. doi: 10.1186/s13047-014-0050-9. eCollection 2014. PMID 25478013